CLINICAL TRIAL: NCT07177664
Title: The Effect of a Nurse Navigation Program on Breastfeeding Self-Efficacy Perception and Breastfeeding Motivation in Primiparous Women: A Randomized Controlled Trial
Brief Title: Effect of a Nurse Navigation Program on Breastfeeding Self-Efficacy and Motivation in Primiparous Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayse Aydin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Fatma OCAKOGLU
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Breastfeeding Education
Keywords: breastfeeding; Breastfeeding Self-Efficacy; Breastfeeding Motivation; Primiparous Women; Nurse Navigation Program; Breastfeeding Counseling
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistics expert, Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Navigation Program Group (Experimental): The study includes women meeting inclusion criteria and consenting to participate. For the randomized intervention group, the process will last about eight months.The first meeting at 28-32 weeks gestation will be at the Family Health Center. The Personal Information Form, Prenatal Breastfeeding Self-Efficacy Scale, and researcher-developed Prenatal Breastfeeding Motivation Checklist will be applied as pretests.Each participant will attend at least four face-to-face sessions-two prenatal and two postpartum-with two additional sessions conducted in person or online per preference.Session 1: 28-32 weeks.
  S2: After 36 weeks, breastfeeding education and brochure; scales repeated.S3: Within one week postpartum; education reinforced; scales applied.S4: 6th postpartum week; training repeated; scales applied S5: 4th postpartum month, face-to-face or online; breastfeeding continuation assessed.S6: 6th postpartum month, face-to-face or online; exclusive breing or complementary feeding assessed.
  Interventions: Other: Breastfeeding Consultation Provided through the Nurse Navigation Program
- Routine Care Group (No Intervention): Data will be collected from the control group at parallel times with the intervention group, which will only receive routine applications without any intervention. In the data collection process, the Personal Information Form, the Prenatal Breastfeeding Self-Efficacy Scale, and the Prenatal Breastfeeding Motivation Table and Breastfeeding Motivation scales developed by the researcher to assess Breastfeeding Motivation will be used in parallel with the intervention group.

INTERVENTIONS:
Other: Breastfeeding Consultation Provided through the Nurse Navigation Program — The navigator nurse will meet with the pregnant woman/mother starting at 28-32 weeks of gestation and continuing until the sixth month postpartum. During these meetings, planned breastfeeding education will be provided, women's questions about breastfeeding will be answered, and counseling will be provided to address any concerns.
  Arms: Nurse Navigation Program Group

SUMMARY:
Objective: To evaluate the effects of a nurse navigation program on breastfeeding self-efficacy and breastfeeding motivation in primiparous women. The research will be conducted as a randomized controlled trial with a pretest-posttest control group.

DETAILED DESCRIPTION:
The study aims to evaluate the effect of a Nurse Navigation Program on breastfeeding self-efficacy perception and breastfeeding motivation in primiparous women. The study population will consist of women aged 18-35 years between the 28th and 32nd weeks of gestation who apply to Yıldızkent, Yenişehir, Adnan Menderes, and Şerif Efendi Family Health Centers between October 2025 and October 2026. Sample size was determined through a priori power analysis using G*Power 3.1.9.4, and repeated measures analysis of variance (ANOVA) was planned. To achieve a power of over 80% at a significance level of 0.05 with a medium effect size, 48 participants were required. Considering potential withdrawal or exclusion, the sample was increased to 100 participants (50 intervention, 50 control). Participants meeting inclusion criteria will be selected by simple random sampling, with allocation to intervention or control groups through randomization. The researcher cannot be blinded, but the statistician will be blinded to group assignment. Data from groups coded as A and B will be analyzed by an independent statistician. The study will follow CONSORT 2010 Flow Diagram guidelines.

Data Collection Data will be collected using the Personal Information Form, Prenatal Breastfeeding Self-Efficacy Scale, Prenatal Breastfeeding Motivation Assessment Checklist, Breastfeeding Self-Efficacy Scale-Short Form, and Primiparous Breastfeeding Motivation Scale. The intervention group will receive structured breastfeeding counseling via the Nurse Navigation Program from the prenatal period until six months postpartum. Scheduled follow-up visits will occur over approximately eight months. The control group will receive routine care only, with data collected in parallel.

Intervention Group

Participants will attend six sessions:

First Meeting: Study orientation, informed consent, baseline assessments including personal information, prenatal self-efficacy, and motivation.

Second Meeting: After 36 weeks, breastfeeding training using a newborn mannequin and educational booklet; post-training reassessment.

Third Meeting: Within seven days postpartum; reinforcement of breastfeeding education and administration of postnatal scales.

Fourth Meeting: End of postpartum 6th week; continued training and scale reassessment.

Fifth Meeting: Fourth postpartum month; conducted online or by phone, infant feeding status assessed.

Sixth Meeting: Sixth postpartum month; online or phone session to evaluate exclusive breastfeeding continuation versus complementary feeding initiation.

Control Group Participants will attend six assessment points corresponding to the intervention group but will receive routine care only. Assessments will be conducted face-to-face, via home visits, or online depending on participant preference.

Data Analysis Data will be coded and analyzed using SPSS version 25. Descriptive statistics will include frequency, percentage, mean, and standard deviation. Normality will be evaluated using skewness and kurtosis coefficients. Appropriate statistical tests will be applied based on data type, including Chi-square, independent samples t-test, Mann-Whitney U, ANOVA, Kruskal-Wallis, paired t-test, Wilcoxon, or Friedman tests. Significance level is p < 0.05. Internal consistency of scales will be assessed with Cronbach's alpha, and effect sizes calculated using Cohen's d or eta-squared for relevant comparisons. All ethical principles will be strictly observed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Being primiparous,
* Not having a health problem that would prevent breastfeeding,
* Being in the 28th-32nd weeks of pregnancy,
* Being between the ages of 18 and 35,
* Having at least a primary school degree,
* Residing in the city center of Erzurum,
* Not having a hearing or vision problem,
* Not having been diagnosed with a psychiatric illness,
* Being fluent in Turkish,
* Being able to use a telephone,
* Women who voluntarily agreed to participate in the study will be included in the sample.

Exclusion Criteria:

* Having given birth before 37 weeks of gestation,
* Having a health problem requiring the newborn to be in intensive care,
* Having a health problem/birth complication that would prevent breastfeeding during the study period,
* Withdrawal from the study at the woman's request,

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — being in the 28th to 32nd week of pregnancy
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 18 months
  There are 15 questions in this form, prepared by the researchers in line with the literature
Prenatal Breastfeeding Self-Efficacy Scale | 18 months
  Prenatal Breastfeeding Self-Efficacy Scale was originally developed to assess pregnant women's perceptions of breastfeeding self-efficacy during the prenatal period. Its validity and reliability for the Turkish context were confirmed in a subsequent adaptation study, which reported a Cronbach's alpha coefficient of 0.86. The scale comprises 20 items, each rated on a 5-point Likert scale ranging from 1 ('Not at all sure') to 5 ('Completely sure'). It is unidimensional, meaning it has no sub-dimensions, and is evaluated based on the total score. The possible total scores range from 20 to 100, with higher scores indicating a greater sense of breastfeeding self-efficacy.
Prenatal Breastfeeding Motivation Assessment Scale | 18 months
  Prenatal Breastfeeding Motivation Assessment Scale was developed by the researcher in the form of a Visual Analog Scale (VAS). Participants are asked to rate their response to the question, "How confident am I that I will be able to breastfeed my baby successfully after birth?" on a scale from 0 = Not confident at all to 10 = Completely confident.
Breastfeeding Self-Efficacy Scale (Short Form) | 18 months
  The original Breastfeeding Self-Efficacy Scale consists of 33 items. The scale was simplified in 2003, resulting in a 14-item short form, referred to as the 'Breastfeeding Self-Efficacy Scale - Short Form.' The scale was culturally adapted into Turkish, and its psychometric properties were evaluated. To determine validity during the antenatal and postnatal periods, construct validity, linguistic validity, and predictive validity analyses were conducted. This is a 5-point Likert-type scale, with responses ranging from '1 = Not at all confident' to '5 = Always confident.' All items are positively worded. Total scores range from 14 to 70, with higher scores indicating greater breastfeeding self-efficacy. Cronbach's alpha coefficient for the scale is 0.93.
Primiparous Breastfeeding Motivation Scale | 18 months
  The scale is a four-point Likert-type instrument, originally comprising 24 items across five subdimensions. During its original development, Cronbach's alpha coefficients for the subdimensions ranged from 0.56 to 0.89. The scale was subsequently adapted into Turkish, resulting in a 23-item version with five subdimensions, validated for use with primiparous women. Items are rated on a four-point Likert-type scale from '1 = Strongly disagree' to '4 = Strongly agree.' Scores for each subdimension are interpreted separately, with higher scores indicating higher motivation levels, rather than computing a total score. For the Turkish-adapted version, the overall internal consistency, measured by Cronbach's alpha, was 0.88.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe AYDIN, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No